CLINICAL TRIAL: NCT06870422
Title: A Randomized, Four-way Change-over Study to Evaluate the Effect of Moderate Heat, Occlusion, and Moderate Exceise on the Pharmacokinetics and Tolerability of the Esflurbiprofen Topical System in Healthy Volunteers
Brief Title: To Assess the Effect of the Special Condition on the Pharmacokinetics and Tolerability of the Esflurbiprofen Topical System (EFTS) in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); HWI pharma services GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TK-254RX-0104; 2024-513059-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- TK-254RX (Experimental): TK-254RX will be applied with no special condition
  Interventions: Drug: Esflurbiprofen Topical System
- TK-254RX with heat (Experimental): TK-254RX will be applied with moderate heat
  Interventions: Drug: Esflurbiprofen Topical System
- TK-254RX with occlusion (Experimental): TK-254RX will be applied with occlusion
  Interventions: Drug: Esflurbiprofen Topical System
- TK-254RX with exercise (Experimental): TK-254RX will be applied with 3 moderate exercise sessions
  Interventions: Drug: Esflurbiprofen Topical System

INTERVENTIONS:
Drug: Esflurbiprofen Topical System — TK-254RX will be applied for one day

SUMMARY:
This study is a single-center, open-label, single-dose trial performed in a randomized, four-way, change-over design in healthy volunteers. The primary purpose of this study is to evaluate the effect of moderate heat, occlusion, and moderate exercise on pharmacokinetics. The secondary purpose is to characterize the effect of special conditions on the bioavailability and to evaluate patch adhesion and safety of TK-254RX and a residual amount of the patch.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 64 years (inclusive)
* body-mass index (BMI): ≧18.5 kg/m² and ≦ 30.0 kg/m²
* good state of health
* non-smoker or ex-smoker for at least 6 months
* written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

* existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* existing or history of hypertension and/or heart failure
* existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
* existing gastrointestinal diseases or pathological findings, which might interfere with the safety and tolerability of the active ingredient
* history of gastrointestinal bleeding or perforation related to previous NSAID therapy
* active, or history of ulcerative colitis, Crohn's disease, peptic ulceration or gastrointestinal haemorrhage
* existing metabolic, endocrine and/or immunologic diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
* diabetes mellitus
* hyperlipidaemia (LDL > 4.16 mmol/l, HDL < 0.91 mmol/l, triglycerides > 2.28 mmol/l, cholesterol > 6.24 mmol/l)
* history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* presence or history of acute or chronic diseases of the skin (e.g., atopic dermatitis (eczema), neurodermatitis, contact allergy, psoriasis, vitiligo, melanoma, squamous cell carcinoma), any dermatological condition or skin sensitivity which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
* existing or history of bronchial asthma
* known allergic reactions (e.g., bronchospasm, rhinitis, angioedema, or urticaria) to the active ingredients used, to acetylsalicylic acid or other NSAIDs, or to constituents of the pharmaceutical preparations
* history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
* systolic blood pressure < 90 or > 139 mmHg
* diastolic blood pressure < 60 or > 89 mmHg
* heart rate < 50 bpm or > 90 bpm
* QTc interval > 450 ms for men and > 470 ms for women
* laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
* ASAT > 20% ULN, ALAT > 10% ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 µmol/l ULN).
* positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
* vaccination against COVID-19 within the last 4 weeks prior to individual intended IMP application
* skin abnormality (e.g., tattoo (including tattoo that was removed), scar, sunburn, or obvious difference in skin colour), open sores, or excessive hair at the application site
* acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
* history of or current drug or alcohol dependence
* positive alcohol or drug test at screening examination
* regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male or ≥ 12 g pure ethanol for female per day
* subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
* regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
* blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
* participation in a clinical trial with administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
* simultaneous participation in another clinical trial with active ingredients
* regular treatment with any systemically available medication (except sexual and thyroid hormones)
* subjects, who report a frequent occurrence of migraine attacks
* positive pregnancy test at screening examination
* pregnant or lactating women
* female subjects who do not agree to apply highly effective contraceptive methods
* subject is vulnerable such as detained or committed to an institution by a court of law or by legal authorities or close affiliation with the sponsor or the investigational site (e.g., a close relative of the investigator, dependent person (e.g., employee of or student at the investigational site), employee of the sponsor or affiliates)
* subjects suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Assessing the effect of each intervention by Area under the plasma concentration versus time curve over 24 hours (AUC0-24) of S-flurbiprofen | Day 1 to Day 2 for each period
  assessment of the effect of heat, occlusion, and moderate exercise on Test by use of AUC0-24 of S flurbiprofen
Assessing the effect of each intervention by peak plasma concentration (Cmax) of S-flurbiprofen | Day 1 to Day 2 for each period
  assessment of the effect of heat, occlusion, and moderate exercise on Test determined by use of Cmax of S flurbiprofen
Assessing the effect of each intervention by area under the plasma concentration versus time curve from patch application to last measurement time point with a concentration value above lower limit of quantitation (AUC0-tlast) of S-flurbiprofen | Day 1 to Day 4 for each period
  assessment of the effect of heat, occlusion, and moderate exercise on Test determined by use of AUC0-tlast of S flurbiprofen
Assessing the effect of each intervention by area under the plasma concentration versus time curve from patch application to infinity (AUC0-inf) of S-flurbiprofen | Day 1 to Day 4 for each period
  assessment of the effect of heat, occlusion, and moderate exercise on Test determined by use of AUC0-inf of S flurbiprofen

SECONDARY OUTCOMES:
Assessing the effect of each intervention by area under the curve over 24 hours (AUC0-24) | Day 1 to Day 2 for each period
  Characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by AUC0-24 of R-flurbiprofen and metabolites, if applicable
Assessing the effect of each intervention by peak plasma concentration (Cmax) | Day 1 to Day 2 for each period
  Characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Cmax of R-flurbiprofen and metabolites, if applicable
Assessing the effect of each intervention by area under the plasma concentration versus time curve from patch application to last time point with a concentration value above lower limit of quantitation (AUC0-tlast) | Day 1 to Day 4 for each period
  Characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by AUC0-tlast of R-flurbiprofen and metabolites, if applicable
Assessing the effect of each intervention by area under plasma concentration versus time curve from patch application to infinity (AUC0-inf) | Day 1 to Day 4 for each period
  Characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by AUC0-inf of R-flurbiprofen and metabolites, if applicable
Assessing the effect of each intervention by percentage of area under the plasma concentration versus time curve extrapolated to infinity to area under the plasma concentration versus time curve from 0 hour to infinity (AUCexpol%) | Day 1 to Day 4 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by AUCexpol% of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Assessing the effect of each intervention by concentration at the last time point with concentration value above lower limit of quantitation (Clast) | Day 1 to Day 2 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Clast of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Assessing the effect of each intervention by time point to reach peak plasma concentration (Tmax) | Day 1 to Day 4 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Tmax of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Asssessing the effect of each intervention by last time point with concentration value above the lower limit of quantitation (Tlast) | Day 1 to Day 4 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Tlast of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Assessing the effect of each intervention by apparent terminal elimination half-life (T1/2) | Day 1 to Day 4 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by T1/2 of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Assessing the effect of each intervention by apparent terminal elimination rate constant determined by log-linear regression (Lz) | Day 1 to Day 4 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Lz of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Assessing the effect of each intervention by time point before first concentration balue above the lower limit quantitation (Tlag) | Day 1 to Day 2 for each period
  characterisation of the effect of heat, occlusion, and moderate exercise on the bioavailability of Test determined by Tlag of S flurbiprofen as well as R flurbiprofen and their metabolites, if applicable
Characterization of EFTS adhesion | Day 2 for each period
  measuring patch adhesion area by percentage of visually by site staff with remaining patch adhered
Characterization of local tolerability | with in 5 minutes after removal of each patch as well as 12 hours, 24 hours, and 36 hours after removal for each period
  Assessing the local tolerability by using the 8-point dermal response and other effects score according to FDA recommendation
Recording adverse event and serious adverse event | Day 1 to Day 4 for each period
Residual amount | Day 2 for each period
  residual amout of S-flurbiprofen in used patch for each period

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Mainzerhofplatz, Erfurt, Germany

IPD SHARING:
Plan to Share IPD: No